CLINICAL TRIAL: NCT02261116
Title: Does Telmisartan Compared to Candesartan Due to a Distinctly Larger Volume of Distribution Exert Stronger Effects in Relevant Peripheral Tissues, e.g. Renal and Adrenal Tissues
Brief Title: Study to Assess Potential Different Properties of Telmisartan Compared to Candesartan in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 502.402
Record Dates: First submitted 2014-10-09; First posted 2014-10-10 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Telmisartan; candesartan; candesartan cilexetil

ARMS (3):
- Telmisartan (Experimental)
  Interventions: Drug: Telmisartan
- Candesartan (Active Comparator)
  Interventions: Drug: Candesartan
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Telmisartan
  Other Names: Micardis®
  Arms: Telmisartan
Drug: Candesartan
  Other Names: Blopress
  Arms: Candesartan
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to assess potential different properties of telmisartan, which due to its Vd, should result in stronger "beneficial" effects of AT1 blockade in tissues (e.g. aldosterone suppression and renin increase) plus stronger AT2 stimulation compared to candesartan

ELIGIBILITY:
Inclusion Criteria:

1. Males, aged 18 to 45 years.
2. Absence of any relevant disease as determined by no clinically deviation from normal in medical history, clinical laboratory determination, ECGs and physical examinations
3. Systolic blood pressure (SBP) between 100 and 140 mmHg systolic and below 85 mmHg diastolic (both left and right arm) and a heart rate of ≥50 bpm
4. Signed informed consent form
5. No intake of drugs inbetween a waiting time of ten times of half-life

Exclusion Criteria:

1. Contraindications to Ang II antagonists, known hypersensitivity, history of angioedema, serious allergy, asthma, allergic skin rash, significant allergic rhinitis or sensitivity to any drug
2. History of cardiovascular diseases: any clinically significant cardio-vascular disease, a supine diastolic blood pressure >86 mmHg and systolic >141 mmHg measured by a standard sphygmomanometer or a heart rate ≤49 bpm
3. Cerebrovascular diseases: history of stroke or transitory ischemic attacks (TIAs) or history of any cerebral bleeding
4. Renal diseases: serum creatinine >1.5 mg/dL
5. Gastrointestinal/Hepatic diseases: Aspartate aminotransferase (ASAT) >40 U/l or Alanine aminotransferase (ALAT) >40 U/L, serum bilirubin >2x upper limit of normal, history of malabsorption or inability to tolerate oral medication, history of gastric or duodenal ulcers, history of significant gastrointestinal bleeding, history of hepatitis within the past years
6. Any history of alcohol or drug abuse
7. Use of any of the following drugs within 4 weeks of study enrolment (e.g. agents known to induce drug metabolizing enzymes): anabolic steroids and corticoids, antiarrhythmics (amiodarone, mexiletine, quinidine, propafenone), antibiotics (chloramphenicol, tetracyclines, sulfonamides, macrolides, cephalosporins, rifampicin, nalidixic acid), antiepileptics (phenytoin, carbamazepine), antifungals (e.g. griseofulvin), barbiturates, cimetidine, ethacrynic acid, fibrates, furosemide, haloperidol, lipid lowering agents (cholestyramine, hydroxymethylglutaryl, coenzyme A (HMG CoA) reductase inhibitors, dextrothyroxin), thyroid replacement therapy hormones or thyrostatics (thioureylene-type). The use of nonsteroidal antiinflammatory drugs (NSAIDs) should be discontinued 2 weeks prior to study enrolment, the one exception of aspirin should be one (1) week prior to study enrolment
8. Participation in any other investigational study, within the 30 days prior to enrolment
9. Blood donation within the previous 3 months
10. The investigator might disqualify a subject for a sound medical or psychiatric reason

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2002-04; Primary Completion 2002-08 (Actual)

PRIMARY OUTCOMES:
Slope of PRA increase versus DR-1 | Predose and 2, 4, 8 h following trial medication
  analysis of variance

SECONDARY OUTCOMES:
Assessment of angiotensin-1 (AT1) pressor antagonism in vivo (DR-1) | Predose and 2, 4, 8 h following trial medication
  rightward shift (DR-1) of diastolic blood pressure response to Angiotensin II dose escalating challenges
Assessment of plasma aldosterone concentration after stimulation with Angiotensin II | Predose and 2, 4, 8 h following trial medication
Reactive response of the plasma renin activity (PRA) | Predose and 2, 4, 8 h following trial medication
Number of subjects with adverse events | up to 42 days